CLINICAL TRIAL: NCT00422409
Title: Palliative Endoscopic Treatment of Malignant GI-strictures With Self Expanding Metal Stents(SEMS)-a Prospective Multicenter Study
Brief Title: Endoscopic Stenting of Gastrointestinal Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ullevaal University Hospital (Other)
Organization: Oslo University Hospital (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 672
Record Dates: First submitted 2007-01-16; First posted 2007-01-17 (Estimated); Last update posted 2011-07-06 (Estimated); Status verified 2007-04

CONDITIONS: Gastrointestinal Neoplasms; Biliary Tract Neoplasms
Keywords: SEMS
MeSH Terms: conditions — Gastrointestinal Neoplasms; Biliary Tract Neoplasms

INTERVENTIONS:
Procedure: Endoscopic stenting

SUMMARY:
Obstruction of the digestive tract is a frequent cause of morbidity in patients with gastrointestinal cancer.Palliative endoscopic treatment with self- expanding metal stents(SEMS)is an alternative to palliative surgery and other palliative treatment options.The method has expanded to include patients with malignancies in the esophagus,gastroduodenal region, biliary tractus and colon. Numerous retrospective studies have reported treatment with SEMS to be safe and effective. Prospective studies,and especially studies regarding Quality of Life improvement are needed.

PURPOSE:

The purpose of this trial is to prospectively study the use and effect of selfexpanding metal stents(SEMS)in a defined population i Norway, especially Quality of Life changes.

DETAILED DESCRIPTION:
The study is divided into four projects:

1. Establish a central register over all patients with malignant GI-obstruction who are treated with SEMS in the Eastern health region in Norway .Treatment incidence, methods used, treatment effect,complications related to the procedure,Need for reinterventions, hospitalisations and survival will be studied.
2. Quality of life(QoL) studies will be performed before and 14 days after treatment.The EORTC QLQ C30 and EORTCs organospecific modules will be used.
3. Gastric emptying before/after stent will be studied.
4. Evaluate SEMS treatment of acute colon obstruction, as a permanent palliative treatment or as a "bridge to surgery"

ELIGIBILITY:
Inclusion Criteria:

* Palliative SEMS treatment for malignant GI-obstruction in esophagus,gastroduodenal region, biliary tractus or colon
* SEMS treatment of acute malignant colon obstruction as a bridge to surgery

Exclusion Criteria:

* Not able to sign informed consent
* SEMS placement in other location last 4 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 270 (Actual)
Dates: Start 2006-10; Primary Completion 2009-04 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Change/improvement i Quality of life

SECONDARY OUTCOMES:
Need for reintervention
Change/improvement in gastric emptying
Rehospitalisations
Complications
Death

CONTACTS AND LOCATIONS:
Overall Officials: Truls Hauge, MD,PhD, Study Director — Ullevaal University Hospital
Locations (7):
- Norway (7):
  - Sentral Hospital Buskerud, Drammen
  - Sentral Hospital Østfold, Fredrikstad
  - Sykehuset Innlandet Gjøvik, Gjøvik
  - Sykehuset Innlandet Lillehammer, Lillehammer
  - Ullevaal University Hospital, Oslo
  - AHUS University Hospital, Oslo
  - Aker University Hospital, Oslo